CLINICAL TRIAL: NCT07131462
Title: Evaluation of Crown Fractures in Permanent Teeth Following Dental Trauma Using the Modified Baysal Dental Trauma Index and Clinical Follow-Up of Their Treatments
Brief Title: Evaluation and Treatment of Crown Fractures Using the Modified Baysal Dental Trauma Index
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Tuba Aydan, Pediatric Dentistry Specialist, Principal Investigator, Inonu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023/69
Record Dates: First submitted 2025-07-29; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Dental Trauma; Crown Fractures; Tooth Fractures
Keywords: Complicated Crown Fractures; Uncomplicated Crown Fractures; Modified Baysal Dental Trauma Index; Permanent Teeth; Pediatric Dentistry
MeSH Terms: conditions — Tooth Fractures | interventions — Endodontics; Dental Pulp Capping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dental Trauma - Crown Fracture Group (Experimental): This arm includes children aged 6 to 14 years who present with crown fractures due to dental trauma. Treatment modality (direct composite restoration, Cvek pulpotomy, or endodontic therapy) will be selected based on clinical and radiographic findings. All patients will be followed over time to assess treatment outcomes.
  Interventions: Procedure: Direct Composite Restoration; Procedure: Cvek Pulpotomy; Procedure: Endodontic Treatment; Procedure: Pulp Capping

INTERVENTIONS:
Procedure: Direct Composite Restoration — Application of direct composite resin to restore the fractured crown of permanent incisors.
Procedure: Cvek Pulpotomy — Partial pulpotomy (Cvek technique) will be performed for complicated crown fractures with vital pulp exposure. The goal is to maintain pulp vitality using biodentin.
Procedure: Endodontic Treatment — Root canal treatment will be applied to teeth with necrotic pulp or extensive pulp exposure not suitable for vital pulp therapy. Procedures will follow standard endodontic protocols.
Procedure: Pulp Capping — In cases of minimal pulp exposure, a direct pulp capping procedure will be performed using biocompatible materials such as calcium hydroxide to preserve pulp vitality.

SUMMARY:
This study will be conducted by the Department of Pediatric Dentistry, Faculty of Dentistry, İnönü University, with the aim of evaluating the treatment processes and follow-up responses of patients aged between 6 and 14 years who will present with crown fractures in their maxillary or mandibular permanent incisors.

Written informed consent will be obtained from the parents of all participating patients. The research will be carried out using a prospective observational design.

Initially, sociodemographic information as well as personal data such as the child's age and gender will be collected through a questionnaire designed for the parents. Additionally, trauma-related information-including the time, location, and cause of the injury-will be recorded in detail using a trauma assessment form developed for the study.

Each patient will undergo clinical and radiographic evaluations, and treatment planning and follow-up will be carried out based on these findings.

DETAILED DESCRIPTION:
The sample size was determined based on a statistical power analysis. This analysis was conducted with an effect size of w = 0.5, an alpha error probability of α = 0.05, and a power of 1 - β = 0.8. Calculations performed for two degrees of freedom (df = 2) yielded a total required sample size of 39 participants.

Inclusion Criteria:

Age between 6 and 14 years Presence of a traumatic dental injury in a permanent tooth Type of TDI classified as either complicated or uncomplicated crown fracture Consent to participate provided by the patient's legal guardian

Exclusion Criteria:

Patients outside the 6-14 age range or presenting for other reasons Patients with traumatic dental injuries other than crown fractures

Types of Treatments Applied for Crown Fractures:

Restoration with composite resin Vital pulp therapies Regeneration Root canal treatment

Clinical Evaluation Criteria of Our Study:

Presence of pain and percussion sensitivity was considered a failure. Presence of abscess and fistula was considered a failure. Repair of the restoration was not considered a failure. Teeth showing loss of vitality and gray discoloration due to necrosis were considered a failure. The treatment success was evaluated using the Periapical Index (PAI) on periapical radiographs obtained from patients included in the study during follow-up visits. Internal and external root resorption were considered failures.

If the radiolucent area observed at the apex had developed or increased after treatment, it was considered a failure.

Reduction of initial radiolucencies observed in baseline radiographs of patients at the start of treatment or in those presenting late was considered a success.

Evaluation was performed according to the Periapical Index (PAI) described by Ørstavik et al. in 1986.

Disruption in the continuity of the lamina dura was considered a failure, whereas formation and continued development of the lamina dura were considered a success.

An increase in root length was considered a success. Calcification observed within the root canals was considered a failure. For immature traumatic teeth with an open apex at the start of treatment, continued and completed root maturation was considered a success.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 14 years
* Presence of traumatic dental injury involving a permanent tooth
* Type of injury classified as a complicated or uncomplicated crown fracture
* Informed consent obtained from the patient's parent or legal guardian

Exclusion Criteria:

* Patients younger than 6 or older than 14 years, or those presenting for non-trauma-related dental issues
* Patients with traumatic dental injuries other than crown fractures (e.g., luxation, avulsion)

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Treated Teeth Without Clinical Symptoms or Radiographic Pathology at 12 Months (PAI Score ≤ 2) | 12 months
  Treatment success will be defined as the absence of spontaneous pain, swelling, sinus tract, abnormal mobility, discoloration, and the presence of radiographic healing or absence of periapical pathology, as assessed using the Periapical Index (PAI) by Ørstavik et al. (1986). Evaluations will be performed at 12 months post-treatment.

SECONDARY OUTCOMES:
Change in Periapical Index (PAI) Score From Baseline to 12 Months | 12 months
  Radiographic healing will be evaluated using the PAI scoring system, comparing baseline and 12-month follow-up periapical radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Aydan, Pediatric Dentistry Specialist, Principal Investigator — Inonu University Faculty of Dentistry
Locations (1):
- Inonu University Faculty of Dentistry, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-29): https://cdn.clinicaltrials.gov/large-docs/62/NCT07131462/Prot_SAP_000.pdf